CLINICAL TRIAL: NCT01005303
Title: A Trial of Micronutrient Supplementation in Patients With Heart Failure
Brief Title: Micronutrient Supplementation in Patients With Heart Failure
Acronym: MINT-HF
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Belfast Health and Social Care Trust (Other)
Responsible Party: Principal Investigator, Pascal McKeown, Principal Investigator, Belfast Health and Social Care Trust
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RGHT000395
Record Dates: First submitted 2009-10-29; First posted 2009-10-30 (Estimated); Results first posted 2023-12-01 (Actual); Last update posted 2023-12-01 (Actual); Status verified 2023-02

CONDITIONS: Heart Failure
Keywords: Heart Failure; Micronutrients; Vitamin D; Inflammation; Oxidative Stress; Quality of Life; Physical Functioning
MeSH Terms: conditions — Heart Failure; Inflammation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Micronutrient (Active Comparator)
  Interventions: Drug: Forceval plus 50 micrograms Vitamin D3

INTERVENTIONS:
Drug: Placebo — 1 Tablet Daily
  Arms: Placebo
Drug: Forceval plus 50 micrograms Vitamin D3 — Forceval: 1 Tablet Daily; Vitamin D3: 2 Tablets Daily
  Arms: Micronutrient

SUMMARY:
There is some evidence to suggest that patients with heart failure may have a reduced dietary intake of vitamins and essential minerals (micronutrients) and that this may worsen the function of the heart. This study is designed to investigate if supplementation with micronutrients (including high-dose vitamin D) will improve the function of the heart in patients with heart failure.

ELIGIBILITY:
Inclusion Criteria:

* New York Heart Association Class II and III
* Already on or tried on best known medical treatment (ACE inhibitor and beta-blocker)
* Stable for a period of at least 6 weeks
* Left ventricular ejection fraction less than or equal to 45%

Exclusion Criteria:

* History of significant alcohol ingestion (more than 40 units per week)
* Severe renal dysfunction (GFR less than 30ml/min)
* Severe hepatic dysfunction (known liver disease or transaminases greater than 3 times the upper limit of normal)
* Atrial fibrillation (in the absence of a pacemaker)
* Frequent ventricular ectopics
* On waiting list for cardiac transplantation
* Uncontrolled diabetes mellitus
* Inability to give informed consent
* Estimated life span less than 12 months
* Already taking a multivitamin/mineral supplement
* Already taking a vitamin-D containing fish oil
* Woman of child-bearing potential
* History of renal stones, hypercalcaemia, sarcoidosis, haemochromatosis or lactose intolerance

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2009-02; Primary Completion 2013-08 (Actual); Study Completion 2015-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pascal McKeown, MD, Principal Investigator — Belfast Health and Social Care Trust; Mark Harbinson, MD, Study Director — Belfast Health and Socail Care Trust; Michelle McKinley, PhD, Study Director — The Queen's Univeristy of Belfast
Locations (1):
- Royal Victoria Hospital, Belfast, United Kingdom

REFERENCES:
- [Derived] McKeag NA, McKinley MC, Harbinson MT, Noad RL, Dixon LH, McGinty A, Neville CE, Woodside JV, McKeown PP. The effect of multiple micronutrient supplementation on left ventricular ejection fraction in patients with chronic stable heart failure: a randomized, placebo-controlled trial. JACC Heart Fail. 2014 Jun;2(3):308-17. doi: 10.1016/j.jchf.2013.12.008. PMID 24952700

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo | Micronutrient
Started | 36 | 38
Completed | 36 | 35 (3 patients did not complete the study protocol (2 developed illnesses during the first 3 months of follow-up, requiring withdrawal from the study, and 1 died approximately 6 months into the study).)
Not Completed | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Micronutrient | Total
Number analyzed (Participants) | 36 | 38 | 74
Age, Continuous [Mean (Standard Deviation); unit: Years] | 62.7 (9.0) | 65.8 (9.4) | 64.3 (9.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 7 | 14
  Male | 29 | 31 | 60
Left Ventricular Ejection Fraction [Mean (Standard Deviation); unit: percentage of LVEF] | 45.1 (9.0) | 38.3 (11.4) | 41.6 (10.8)
New York Heart Association Functional Class II [Count of Participants; unit: Participants] — New York Heart Association Functional Class II = Slight limitation of physical activity. Comfortable at rest. Ordinary physical activity results in fatigue, palpitation, dyspnea (shortness of breath). This was assessed via clinical history.
  Participants | 30 | 28 | 58
New York Heart Association Functional Class III [Count of Participants; unit: Participants] — New York Heart Association Functional Class III = Marked limitation of physical activity. Comfortable at rest. Less than ordinary activity causes fatigue, palpitation, or dyspnea.This was assessed via clinical history.
  Participants | 6 | 10 | 16
Aetiology Ischaemic [Count of Participants; unit: Participants] | 19 | 28 | 47
Aetiology Non-Ischaemic [Count of Participants; unit: Participants] | 17 | 10 | 27
Angiotensin Converting Enzyme inhibitor or Angiotensin Receptor Blocker [Count of Participants; unit: Participants] | 36 | 36 | 72
Beta-Blocker [Count of Participants; unit: Participants] | 34 | 36 | 70
Mineralocorticoid Receptor Antagonist [Count of Participants; unit: Participants] | 13 | 24 | 37
Implantable Cardioverter Defibrillator [Count of Participants; unit: Participants] | 18 | 24 | 42
Cardiac Resynchronisation Therapy [Count of Participants; unit: Participants] | 10 | 12 | 22

OUTCOME MEASURES:

1. Primary Outcome: Left Ventricular Ejection Fraction
Time Frame: Baseline, and 12 months
Population: Result not available for 3 patients: 1 patient was unable to attend for 12 month scan due to personal reasons, 1 patient was unable to attend due to illness and images from 1 patient of inadequate quality for analysis.
Measure: Mean (Standard Deviation); unit: percentage of LVEF
Arm/Group | Placebo | Micronutrient
Number analyzed (Participants) | 35 | 33
percentage of LVEF
  Baseline | 44.7 (8.8) | 38.9 (11.1)
  12 months | 44.9 (12.0) | 38.6 (10.9)

2. Secondary Outcome: Quality of Life Questionnaire Score
Description: Minnesota Living With Heart Failure Questionnaire. The questionnaire is comprised of 21 questions around several physical, emotional and socioeconomic ways heart failure can adversely affect a patient's life. After receiving brief standardized instructions, the patient marks a 0 (zero) to 5 (five) scale to indicate the extent to which each itemized adversity of heart failure has prevented the patient from living as they wanted to live during the past 4 weeks. The questionnaire is simply scored by summation of all 21 responses (score range 0-105). Higher scores indicate worse quality of life.
Time Frame: Baseline, and 12 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Micronutrient
Number analyzed (Participants) | 36 | 35
units on a scale
  Baseline | 33.7 (25.2) | 34.0 (22.6)
  12 months | 38.2 (24.1) | 33.1 (21.6)

3. Secondary Outcome: Six Minute Walk Test Distance
Time Frame: Baseline, and 12 months
Population: Result not available for 6 patients: all were unable to perform six minute walk test due to joint disease / poor mobility.
Measure: Mean (Standard Deviation); unit: Metres
Arm/Group | Placebo | Micronutrient
Number analyzed (Participants) | 33 | 33
Metres
  Baseline | 437.8 (94.9) | 417.0 (120.1)
  12 months | 440.2 (98.6) | 412.5 (114.9)

4. Secondary Outcome: Serum N-terminal Prohormone of Brain Natriuretic Peptide (NT-proBNP) Concentration
Time Frame: Baseline, and 12 months
Measure: Mean (Standard Deviation); unit: ng/L
Arm/Group | Placebo | Micronutrient
Number analyzed (Participants) | 36 | 35
ng/L
  Baseline | 841.6 (1137.9) | 1293.4 (2064.1)
  12 months | 1343.6 (2983.7) | 1763.6 (5024.5)

5. Secondary Outcome: Serum C-reactive Protein (CRP) Concentration
Time Frame: Baseline, and 12 months
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Placebo | Micronutrient
Number analyzed (Participants) | 36 | 35
mg/L
  Baseline | 5.6 (8.7) | 6.3 (15.0)
  12 months | 4.3 (3.8) | 4.6 (5.4)

6. Secondary Outcome: Serum Tumor Necrosis Factor-alpha (TNF-α) Concentration
Time Frame: Baseline, and 12 months
Population: Result not available for 3 patients: all due to quality control (intra-assay coefficient of variation > 25%).
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Placebo | Micronutrient
Number analyzed (Participants) | 33 | 35
pg/mL
  Baseline | 4.4 (1.5) | 4.1 (1.3)
  12 months | 4.6 (1.6) | 4.1 (1.4)

7. Secondary Outcome: Serum Interleukin-6 (IL-6) Concentration
Time Frame: Baseline, and 12 months
Population: Result not available for 5 patients: all due to quality control (intra-assay coefficient of variation > 25%).
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Placebo | Micronutrient
Number analyzed (Participants) | 32 | 34
pg/mL
  Baseline | 5.0 (6.5) | 7.1 (12.5)
  12 months | 5.0 (6.3) | 4.2 (3.8)

8. Secondary Outcome: Serum Interleukin-10 (IL-10) Concentration
Time Frame: Baseline, and 12 months
Population: Result not available for 10 patients: all due to due to quality control (intra-assay coefficient of variation > 25%).
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Placebo | Micronutrient
Number analyzed (Participants) | 34 | 27
pg/mL
  Baseline | 1.5 (2.1) | 1.2 (0.7)
  12 months | 1.5 (1.5) | 1.1 (0.5)

9. Secondary Outcome: Urinary 8-iso-prostaglandin F2 Alpha (8-iso-PGF2α) Concentration
Time Frame: Baseline, and 12 months
Measure: Mean (Standard Deviation); unit: mol/mmol creatinine
Arm/Group | Placebo | Micronutrient
Number analyzed (Participants) | 36 | 35
mol/mmol creatinine
  Baseline | 11.3 (5.8) | 12.1 (7.2)
  12 months | 11.7 (4.6) | 10.5 (3.8)

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | Placebo | Micronutrient
All-Cause Mortality (participants affected / at risk) | 0/36 | 1/38
Serious Adverse Events (participants affected / at risk) | 18/36 | 10/38
Other Adverse Events (participants affected / at risk) | 0/36 | 0/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=36) | Micronutrient (N=38)
Hospital Admission (Cardiac disorders) | 18 | 10 — Hospital admission for any reason

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes